CLINICAL TRIAL: NCT00384826
Title: Effect of an Early Therapeutic Permutation on the Tumoral Control of Patients Receiving in First Line a Specific Inhibitor of Tyrosin Kinase of EGFR (Erlotinib) or a Taxan-based Chemotherapy for the Treatment of Not Resecable Adenocarcinoma With Bronchiolo-alveolar.
Brief Title: Therapeutic Strategy in Advanced Bronchioloalveolar Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-0504
Record Dates: First submitted 2006-10-05; First posted 2006-10-06 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Adenocarcinoma, Bronchiolo-Alveolar
Keywords: Adenocarcinoma, Bronchiolo-Alveolar
MeSH Terms: conditions — Adenocarcinoma, Bronchiolo-Alveolar | interventions — Erlotinib Hydrochloride; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: erlotinib
- 2 (Experimental)
  Interventions: Drug: paclitaxel + carboplatine

INTERVENTIONS:
Drug: erlotinib — Erlotinib 150 mg/day (until progression)
  Arms: 1
Drug: paclitaxel + carboplatine — Paclitaxel 90 mg/m² D1, D8, D15 (D1=D28, until progression) Carboplatine AUC 6 D1 (D1=D28, 6 cycles)
  Arms: 2

SUMMARY:
To evaluate among patients with untreated advanced ADC-CBA, impact on the disease control rate after 4 months treatment of an early therapeutic permutation with the first month in the absence of stabilization or objective answer.

ELIGIBILITY:
Inclusion Criteria:

* CBA histologically proven (or cytologically with pneumonic presentation) PS < 3 signed and written informed consent

Exclusion Criteria:

* visible tumoral lesion in bronchial fibroscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2006-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
16-week Disease Control Rate | 4-week

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Cadranel, Principal Investigator — APHP Hopital Tenon (Pneumologie) - Paris - France
Locations (9):
- France (9):
  - Centre Hospitalier - Pneumologie, Belfort
  - APHP - CHU Avicenne - Oncologie Medicale, Bobigny
  - Centre F. Baclesse, Caen
  - CHU - Pneumologie, Caen
  - CHU Grenoble - pneumologie, Grenoble
  - APHP - Saint-Antoine - pneumologie, Paris
  - APHP - Hopital Tenon - Pneumologie, Paris
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - CHU Lyautey - Pneumologie, Strasbourg

REFERENCES:
- [Background] Wislez M, Gounant V, Cadranel J. [Bronchioloalveolar carcinoma]. Rev Mal Respir. 2005 Dec;22(6 Pt 2):8S70-5. French. PMID 16340839
- [Background] Wislez M, Massiani MA, Milleron B, Souidi A, Carette MF, Antoine M, Cadranel J. Clinical characteristics of pneumonic-type adenocarcinoma of the lung. Chest. 2003 Jun;123(6):1868-77. doi: 10.1378/chest.123.6.1868. PMID 12796162
- [Derived] Cadranel J, Gervais R, Merle P, Moro-Sibilot D, Westeel V, Bigay-Game L, Quoix E, Friard S, Barlesi F, Lethrosne C, Moreau L, Monnet I, Salaun M, Oliviero G, Souquet PJ, Antoine M, Langlais A, Morin F, Wislez M, Zalcman G; Intergroupe Francophone de Cancerologie Thoracique (IFCT). Erlotinib versus carboplatin and paclitaxel in advanced lepidic adenocarcinoma: IFCT-0504. Eur Respir J. 2015 Nov;46(5):1440-50. doi: 10.1183/13993003.02358-2014. Epub 2015 Sep 17. PMID 26381515
- See also: Official French Intergroup website — http://www.ifct.fr